CLINICAL TRIAL: NCT05582265
Title: A Phase 3, Prospective，Multicenter, Randomized Open-Label Trial to Compare the Efficacy and Safety of Tislelizumab (BGB A317, Anti-PD1 Antibody) Combined With Chemotherapy Followed By Surgery Versus Up-Front Surgery as Treatment for Resectable Head And Neck Squamous Cell Carcinoma
Brief Title: Tislelizumab Combined With Chemotherapy Followed by Surgery Versus Up-front Surgery in Resectable Head and Neck Squamous Cell Carcinoma (REDUCTION-I)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Zhongshan People's Hospital, Guangdong, China (Other); Shenzhen Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Song Fan, MD, Associate Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2022-256-1
Record Dates: First submitted 2022-10-11; First posted 2022-10-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Head and Neck Squamous Cell Carcinomas
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiation; Carboplatin; Neoadjuvant Therapy; Adjuvants, Pharmaceutic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neoadjuvant Tislelizumab + Reduction of Cycles of Chemotherapy (Arm A) (Experimental): Neoadjuvant therapy ( 3 cycles ) ： Cycle1（Cycle length: 21 days）：Tislelizumab (IV), dose= 200mg, day=1; Cisplatin (IV), dose=75 mg/m2, or Carboplatin (IV), AUC=5, day=1; Nab-paclitaxel (IV), dose=260mg/m2, day=1.
  Cycle2、3（Cycle length: 21 days）：Tislelizumab (IV), dose= 200mg, day=1.
  Following surgical resection, high risk participants receive 200 mg Tislelizumab Q3W plus chemoradiotherapy as adjuvant therapy. Low risk participants receive 200 mg Tislelizumab Q3W plus radiotherapy as adjuvant therapy.
  Interventions: Drug: Tislelizumab（neoadjuvant）; Drug: Cisplatin （neoadjuvant）; Drug: Nab-paclitaxel （neoadjuvant）; Procedure: Surgical resection; Drug: Cisplatin（adjuvant）; Drug: Tislelizumab（adjuvant）; Radiation: Radiation; Drug: Carboplatin (neoadjuvant）; Drug: Carboplatin (adjuvant）
- Neoadjuvant Tislelizumab + Chemotherapy (Arm B) (Experimental): Neoadjuvant therapy ( 3 cycles ) ： Cycle1、2、3（Cycle length: 21 days）：Tislelizumab (IV), dose= 200mg, day=1; Cisplatin (IV), dose=75 mg/m2, or Carboplatin (IV), AUC=5, day=1; Nab-paclitaxel (IV), dose=260mg/m2, day=1.
  Following surgical resection, high risk participants receive 200 mg Tislelizumab Q3W plus chemoradiotherapy as adjuvant therapy. Low risk participants receive 200 mg Tislelizumab Q3W plus radiotherapy as adjuvant therapy.
  Interventions: Drug: Tislelizumab（neoadjuvant）; Drug: Cisplatin （neoadjuvant）; Drug: Nab-paclitaxel （neoadjuvant）; Procedure: Surgical resection; Drug: Cisplatin（adjuvant）; Drug: Tislelizumab（adjuvant）; Radiation: Radiation; Drug: Carboplatin (neoadjuvant）; Drug: Carboplatin (adjuvant）
- Up-front Surgery (Arm C) (Other): Following surgical resection, high risk participants receive chemoradiotherapy as adjuvant therapy. Low risk participants receive radiotherapy as adjuvant therapy.
  Interventions: Procedure: Surgical resection; Drug: Cisplatin（adjuvant）; Radiation: Radiation; Drug: Carboplatin (adjuvant）

INTERVENTIONS:
Drug: Tislelizumab（neoadjuvant） — Tislelizumab 200 mg administered by intravenous (IV) infusion on Day 1 of each 21-day cycle
  Arms: Neoadjuvant Tislelizumab + Chemotherapy (Arm B); Neoadjuvant Tislelizumab + Reduction of Cycles of Chemotherapy (Arm A)
Drug: Cisplatin （neoadjuvant） — Cisplatin 75 mg/m2 administered by intravenous (IV) infusion on Day 1 of each 21-day cycle
  Arms: Neoadjuvant Tislelizumab + Chemotherapy (Arm B); Neoadjuvant Tislelizumab + Reduction of Cycles of Chemotherapy (Arm A)
Drug: Nab-paclitaxel （neoadjuvant） — Nab-paclitaxel 260mg/m2 administered by intravenous (IV) infusion on Day 1 of each 21-day cycle
  Arms: Neoadjuvant Tislelizumab + Chemotherapy (Arm B); Neoadjuvant Tislelizumab + Reduction of Cycles of Chemotherapy (Arm A)
Procedure: Surgical resection — Standard of care
Drug: Cisplatin（adjuvant） — Cisplatin 100 mg/m2 administered by intravenous (IV) infusion on Day 1 of each 21-day cycle
Drug: Tislelizumab（adjuvant） — Tislelizumab 200 mg administered by intravenous (IV) infusion on Day 1 of each 21-day cycle
  Arms: Neoadjuvant Tislelizumab + Chemotherapy (Arm B); Neoadjuvant Tislelizumab + Reduction of Cycles of Chemotherapy (Arm A)
Radiation: Radiation — Recommended, standard of care
Drug: Carboplatin (neoadjuvant） — Carboplatin (IV), AUC=5，administered by intravenous (IV) infusion on Day 1 of each 21-day cycle
  Arms: Neoadjuvant Tislelizumab + Chemotherapy (Arm B); Neoadjuvant Tislelizumab + Reduction of Cycles of Chemotherapy (Arm A)
Drug: Carboplatin (adjuvant） — Carboplatin (IV), AUC=5，administered by intravenous (IV) infusion on Day 1 of each 21-day cycle

SUMMARY:
A prospective, randomized, open-label, multicenter Phase 3 trial designed to compare the safety and efficacy of Tislelizumab combined with chemotherapy followed by surgery versus up-front surgery in resectable head and neck squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

Have a histologically confirmed diagnosis of HNSCC which is planned for treatment with curative intent including surgical resection: stage III/IVA.

Greater than or equal to 18 and less than 80 years of age at time of study entry.

ECOG performance status of 0 or 1. Measurable disease as per RECIST 1.1. Patients must have no prior exposure to immune-mediated therapy, including anti- cytotoxic T-lymphocyte protein 4 (CTLA-4), anti-programmed cell death 1, anti-programmed cell death 1 ligand 1 (PD-L1), or anti-programmed cell death ligand 2 antibodies, excluding therapeutic anticancer vaccines.

Screening labs must meet the following criteria and must be obtained within 14 days prior to registration:

Adequate hepatic and renal function as demonstrated by

Serum creatinine < 1.5 X ULN or CrCl > 40mL/min (if using the Cockcroft-Gault formula below):

Males: Creatinine CL (mL/min) = (Weight (kg) x (140 - Age))/(72 x serum creatinine (mg/dL)） Females: Creatinine CL (mL/min) = (Weight (kg) x (140 - Age))/(72 x serum creatinine (mg/dL))x 0.85 AST/ALT ≤ 3 x ULN Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)

Adequate bone marrow function as demonstrated by:

Absolute Neutrophil Count >1,500/µL Platelets > 100 X 103/µL Hemoglobin > 9.0 g/dL Women of reproductive potential should have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 21 days of study enrollment.

Women of reproductive potential must use highly effective contraception methods to avoid pregnancy for 23 weeks after the last dose of study drugs; "women of reproductive potential" is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal; menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes; in addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL.

Men of reproductive potential who are sexually active with women of reproductive potential must use any contraceptive method with a failure rate of less than 1% per year; men who are receiving the study medications will be instructed to adhere to contraception for 31 weeks after the last dose of study drugs; men who are azoospermic do not require contraception.

Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Subjects must agree to allow use of any pre-treatment tissue remaining after definitive diagnosis is made (ie, archival and or fresh tissue) for research purposes. In addition, subjects must consent to allow use of their residual post-operative tissue for research purposes.

Exclusion Criteria:

Is currently participating in or has participated in a study of an investigational agent within 4 weeks of the first dose of treatment or has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.

Has had another known invasive malignancy within the previous 5 years and/or has had surgery, chemotherapy, targeted small molecule therapy or radiation therapy within 5 years for a known malignancy prior to study day 0.

If subject received major surgery for any other reason, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.

Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of day -5. Inhaled or topical steroids, and adrenal replacement steroid > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.

Has an active autoimmune disease requiring systemic steroid treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids.

Active, known or suspected autoimmune disease. Note: Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger .

Has evidence of interstitial lung disease or active, non-infectious pneumonitis.

Has an active infection requiring systemic therapy. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways.

A history of allergic reaction attributed to compounds of similar chemical or biologic composition to the treatment or other agents used in the study.

Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 23 weeks after the last dose of trial treatment.

Has a known history of Human Immunodeficiency Virus (HIV) infection (HIV 1/2 antibodies).

Has known active Hepatitis B or C. Known history of active TB (bacillus tuberculosis ).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 537 (Estimated)
Dates: Start 2022-10-28 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Event-free Survival (EFS) | Up to 3 years
  EFS is the time from the date of randomization to the date of first record of any of the following events: disease progression; local or distant recurrence as assessed with imaging or biopsy as indicated; or death due to any cause.

SECONDARY OUTCOMES:
Percentage of Participants Who Experienced High-Grade (Grade 3-4 and Grade 5) Adverse Events | From time of first dose of study treatment until the end of follow-up (up to 5 years)
  High-grade adverse events were tabulated using worst grade per Common Terminology Criteria for Adverse Events, National Cancer Institute (NCI CTCAE) Version 5.0 criteria.
Pathological complete response (pCR) rate | Up to 30 days post-sugery
  pCR is defined as the absence of invasive squamous cell carcinoma within the resected primary tumor specimen and all the sampled regional lymph nodes.
Major Pathological Response (MPR) rate | Up to 30 days post-sugery
  MPR is defined as ≤10% invasive squamous cell carcinoma within the resected primary tumor specimen and all the sampled regional lymph nodes.
Event-free Survival (EFS) | Up to 5 years
  EFS is the time from the date of randomization to the date of first record of any of the following events: disease progression; local or distant recurrence as assessed with imaging or biopsy as indicated; or death due to any cause.
Objective Response Rate (ORR) | Up to 30 days post-sugery
  The rate of patients with complete remission (CR) or partial response (PR) evaluated by RECIST 1.1 criteria by site radiology review.

OTHER OUTCOMES:
Percentage of Participants Experiencing An Adverse Event (AEs) | From time of first dose of study treatment until the end of follow-up (up to 5 years)
  Percentage of adverse events that are possibly, probably or definitely related to study treatment per Criteria for Adverse Events version 5 (CTCAE v5.0).
Event-free Survival (EFS) | Up to 3 years
  EFS is the time from the date of randomization to the date of first record of any of the following events: disease progression; local or distant recurrence as assessed with imaging or biopsy as indicated; or death due to any cause（Arm A versus Arm B）.

CONTACTS AND LOCATIONS:
Overall Officials: Song Fan, Doctor, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (3):
- China (3):
  - Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guanzhou, Guangdong
  - Zhong shan people's hospital, Zhongshan, Guangdong
  - Huazhong University of Science and Technology Union Hospital (Nanshan Hospital), Shenzhen, Nanshan